CLINICAL TRIAL: NCT06497400
Title: Pilot Randomized Controlled Trial of Brazilian Jiu Jitsu (BJJ) Training Versus Hatha Yoga for Symptoms of Post-Traumatic Stress Disorder (PTSD) Among U.S. Male Veterans
Brief Title: Brazilian Jiu Jitsu vs. Yoga for Treating Symptoms of PTSD
Acronym: JOYPTSDVET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Responsible Party: Principal Investigator, Alison Willing, Professor, University of South Florida
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 00026323
Record Dates: First submitted 2019-04-19; First posted 2024-07-11 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Post Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Waiting Lists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Brazilian Jiu Jitsu (Active Comparator): Jiu Jitsu intervention for ten weeks
  Interventions: Other: Brazilian Jiu Jitsu
- Hatha Yoga (Active Comparator): Yoga intervention for ten weeks
  Interventions: Other: Hatha Yoga
- Waitlist (Active Comparator): Waitlist group for 5 weeks, then allowed to chose if they want to be in Group A Jiu Jitsu or Group B Yoga for ten week intervention
  Interventions: Other: Waitlist

INTERVENTIONS:
Other: Brazilian Jiu Jitsu — Instruction of two classes each week for ten weeks of Brazilian Jiu Jitsu
  Arms: Brazilian Jiu Jitsu
Other: Hatha Yoga — Instruction of two classes each week for ten weeks of Hatha Yoga
  Arms: Hatha Yoga
Other: Waitlist — Participant will waitlist for 5 weeks and then be allowed to decide which intervention they want to do Group A/ Jiu Jitsu or Group B/Yoga for ten weeks..
  Arms: Waitlist

SUMMARY:
Post-traumatic stress disorder (PTSD) is a disabling anxiety disorder that may occur after witnessing a traumatic event, and that evokes a combination of intrusion and avoidance symptoms, negative alterations in cognitions and mood, and alterations in arousal and reactivity1.

The primary objective of this pilot randomized controlled trial is to estimate and compare the effects of the practice of Brazilian Jiu Jitsu (BJJ) vs. hatha yoga vs. a waitlist control condition in influencing symptoms of PTSD, related comorbidities, post-traumatic growth, and quality of life among U.S. service members/veterans with current symptoms of PTSD. In addition, objective measurements (comparisons) of stress and sleep quality will be made through the collection and evaluation of salivary alpha amylase, hair cortisol, and actigraphy, a non-invasive way to measure activity cycles.

DETAILED DESCRIPTION:
The design is a three arm randomized controlled pilot trial comparing the effects of a 10-week BJJ program (n=10) and a 10-week hatha yoga program (n=10) vs. a 5-week waitlist control regimen (n=5). Subjects randomly assigned to the waitlist condition will be offered the choice of participating in the BJJ or yoga intervention after the 5-week waitlist period. By trial inclusion criteria, all subjects will be male U.S. service members or veterans who report significant symptoms of PTSD (as determined by the 20-item PTSD checklist (PCL-5) and supplemental measures. Assessments will occur pre-intervention, at the midpoint of the intervention (5 weeks), at the end of the assigned intervention period (10 weeks), and at 2-month follow-up for the BJJ and yoga arms of the trial. Study variables will consist of reliable and valid self-report measures of symptom status to be completed by all study participants. In addition, saliva samples will be collected before and after individual sessions of BJJ/Yoga at 3 timepoints: first session, mid-point session at 5 weeks, and final session at 10 weeks. The same measurement schedule will be used for collection of hair cortisol samples and actigraphy assessment of sleep quality captured from wearing a watch for a one-week period of time at baseline, 5-weeks, and 10-weeks. The waitlist control group will wear the actigraphy watch at baseline and 5 weeks.

The trial will estimate effect size of the 2 active treatment arms (BJJ, Yoga) compared to the waitlist condition, and similarly, examine whether the BJJ arm appears to be non-inferior to the Yoga arm of the trial. Whereas the trial, designed as a pilot, is not powered for formal hypothesis testing, estimates of effect size will be examined with respect to the following underlying hypotheses:

1. Both the BJJ and Hatha Yoga regimens will provide evidence suggestive of superiority compared to the waitlist control regimen with respect to the primary outcome of symptoms of PTSD, as well as secondary outcomes.
2. Results will provide evidence suggestive of non-inferiority of the BJJ regimen compared to Hatha Yoga with respect to the primary outcome of symptoms of PTSD, as well as secondary outcomes.

Analyses will inform the design of a future planned large clinical trial to determine the potential benefit of BJJ and/or Yoga in reducing symptoms of PTSD and related comorbidities.

ELIGIBILITY:
Inclusion Criteria:

* Male U.S. service member or veteran
* Current evidence of significant symptoms of PTSD, indicative of probable diagnosis of PTSD, as determined from the 20-item PCL-5, and positive screen on the PTSD subscale of the Psychiatric Diagnostic Screening Questionnaire (PDSQ)
* Denial of suicidal/homicidal ideation or intent, and no evidence of psychotic behavior or being in psychological crisis
* Ability to read and speak English
* between 18 - 44 years of age or older

Exclusion Criteria:

* Previous enrollment (past 6 months) in JJ regimen or Yoga regimen consistent with the regimens to be provided as the study interventions
* Major psychiatric disorder (e.g. bipolar disorder) uncontrolled and likely to interfere with treatment delivery (as determined by clinician assessment)
* Current substance abuse dependence (alcohol and/or drug) treatment anticipated to interfere with treatment delivery (i.e. exhibiting significant withdrawal symptoms or inability to refrain from substance dependence immediately prior to intervention sessions).
* Brain injury prohibiting speech, writing, and purposeful actions or screen positive for traumatic brain injury (history of concussion is acceptable).
* Cognitive impairment that prohibits informed consent and/or compliance to the study protocol.
* Contraindication to significant physical activity with BJJ or Yoga.

Ages: 18 Years to 44 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2017-07-30 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Change in PTSD Checklist - 5 (PCL-5) score | Change from pre-intervention to 2 months after completion of BJJ training
  There are 20 questions that inquire about the different symptoms that correspond to 4 different types of PTSD symptoms (intrusion, avoidances, negative affect and hyperarousal). Each item is scored on a 5-point Likert scale from 0 (hasn't bothered a person in the past 2 weeks) to 4 (bothers the person all the time). We used total score on this test.

SECONDARY OUTCOMES:
Change in Posttraumatic Growth Inventory-Short form (PTGI-SF) | Change from pre-intervention to 2 months after completion of BJJ training
  This scale assesses positive changes that may follow traumatic events. It consists of 10 items scored from "0" to "5" with 0 representing "no experience of change as a result of my crisis" and 5 representing "experiencing the change to a very great degree." The score from each item is summed to give a total score.
Change in Brief Symptom Inventory -18 (BSI-18) score | Change from pre-intervention to 2 months after completion of BJJ training
  This scale is the shortened form of the Symptom Checklist 90-Revised (SCL-90-R). There are 18 items that address clinically relevant psychological symptoms in adolescents and adults that cover three factors - Somatization, Depression, and Anxiety - as well as a Global Severity Index. We used the Global Severity Score which is simply the summation of all the scales. The study subject is asked to score each item from 0 (not at all) to 4 (extremely) with respect to the last 7 days.
Change in score on the Centers for Epidemiological Studies Depression Scale (CES-D) | Change from pre-intervention to 2 months after completion of BJJ training
  The CES-D is a self-report scale that measures depressive symptomatology during the past week. There are 20 items and they are rated depending on whether the statement is worded positively or negatively. For positively worded questions, the scoring is:
  * Most or all of the time (5-7 days) = 0
  * Occasionally or a moderate amount of time (3-4 days) = 1
  * Some or a little of the time (1-2 days) = 2
  * Rarely or none of the time (less than 1 day) = 3.
  For negatively worded questions, the scores are opposite:
  * Most or all of the time (5-7 days) = 3
  * Occasionally or a moderate amount of time (3-4 days) = 2
  * Some or a little of the time (1-2 days) = 1
  * Rarely or none of the time (less than 1 day) = 0
  The scores on each item are simply added together. Total score can range from 0-60.
Change in score on the Pittsburgh Sleep Quality Index (PSQI) | Change from pre-intervention to 2 months after completion of BJJ training
  This self-report scale measures quality and patterns of sleep in adults over the prior month. In the first four questions, the participants are asked to provide discrete answers about bedtime, how long it takes them to fall asleep, what time do they get up in the morning and how many hours they sleep. All remaining questions are scored on a 4-point Likert scale. Standard scoring protocol will be performed. Total score on the test can range from 0-21.
Change in score on the Pain Outcomes Questionnaire - Short Form (POQ) | Change from pre-intervention to 2 months after completion of BJJ training
  This instrument assesses specific aspects of pain on five basic categories that include Activities of Daily Living (ADL), Mobility, Negative Affect (NA), Vitality, and Fear. Each item is scored on a scale of 0-10 with higher scores representing increase severity. Total score was used.
Change in Use of Medications | Change from pre-intervention to 2 months after completion of BJJ training
  This is a self-made form that asks study participants to disclose medications that they are using and if medication use changes over time and with BJJ training
Change in score on the Alcohol Use Disorder Identification Test (AUDIT) | Change from pre-intervention to 2 months after completion of BJJ training
  This instrument assesses alcohol consumption, drinking behaviors, and alcohol-related problems. There are 10 questions that are scored with a Likert scale ranging from "0" (Never) to "4" (4 or more times a week). Scores are totaled over the 10 questions. Total score ranges from 0-40, a score of 8 or more indicating potentially harmful behavior.

CONTACTS AND LOCATIONS:
Locations (1):
- University of South Florida/Center of Excellence for Aging and Brain Repair/department of Neurosurgery, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No